CLINICAL TRIAL: NCT05970952
Title: Incidence, Risk Factors, and Outcomes for Acute Kidney Injury in Intensive Care Patients: a Prospective Observational Study
Brief Title: Acute Kidney Injury in Intensive Care Patients
Acronym: AKI-ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 82-2023
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Acute Renal Injury; Critical Illness
Keywords: acute renal injury; intensive care unit
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational study is to evaluate the incidence, risk factors, and outcomes for development of acute kidney injury (AKI) in intensive care pateints.

The main questions it aims to answer are:

* What is the incidence of acute kidney injury in intensive care patients?
* What are risk factors for development of acute kidney injury? All adult patients admitted to the ICU with a stay of 48 h or more will be included in the study.

DETAILED DESCRIPTION:
Material Methods:

Study design and setting: This study is designed as an prospective observational clinical trial to investigate incidence, causes, risk factors and outcome of AKI in critically ill patients. It will be performed in the medical-surgical ICU with 50 beds of the Health Science University Haseki Research and Training Hospital, a referral hospital with 700 beds in Istanbul, Turkey. It will be carried out according to the Declaration of Helsinki with the approval of the local Institutional Review Board (Date/number: 26 April 2023/82) and informed consent will be obtained from all patients or their family members.

Patients selection: All adult patients admitted to the ICU with a stay of 48 h or more will be included in the study. Patients with missing data, end-stage renal disease, existence of AKI at the time of ICU admission or history of renal transplantation will be excluded from the study. Patients that were readmitted to the ICU within 48 h will reunited with the first admission and be considered as one admission for the analysis. The follow-up period is limited to 28 days.

Data collection: In enrolled patients data on demographic characteristics (age, sex, height, weight, body mass index) will be obtained. Lengths of stay (LOSs) in the ICU and hospital, main reason for ICU admittance, co-morbid conditions, organ failures developed during ICU stay and presence of contrast exposure will be recorded as well as data on mechanical ventilation, renal replacement therapies and invasive procedures including central venous line placement, arterial line placement and tracheostomy. Laboratory test results including blood count, coagulation parameters, blood biochemistry parameters and arterial blood gases will be collected daily along with urine analysis, urinary output and fluid balance. Data on drugs including vasoactive, inotropic, corticosteroid, diuretic, antiinfective agents will be noted daily. Blood and blood components transfusions will also be recorded. Moreover presence and duration of hypotension (mean arterial pressure <70 mmHg) and rhythm disorders will be recorded. Severity of illness will be evaluated by using Acute Physiology and Chronic Health Evaluation (APACHE) II scores at the time of ICU admission.

Outcomes and definitions: The primary outcome variable of the study is to detect the incidence of AKI. The diagnosis and classification of AKI will be performed according to the KDIGO criteria based on changes in serum creatinine (SCr) or urine output.31 If available, SCr value measured within a 3-month period prior to ICU admission will be defined as baseline value. If no such value existed, SCr value at the time of admission to the ICU will be considered as baseline value. CKD will be defined as an estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73m2 computed by using MDRD equation according to the KDIGO recommendations.31 Secondary outcome variables included all-cause mortality, clinical and laboratory risk factors for the development of AKI as described above.

Statistical analysis: Statistical analysis was performed using the SPSS software package for Windows (Statistical Package for Social Sciences, version 22.0; SPSS Inc., Chicago, Illinois, USA). In the power analysis based on previous studies, it was calculated that at least 159 patients should be included in the study for 0.05 type 1 error and 80% power. Descriptive statistics will given as numbers and percentages for categorical variables or as the mean ± standard deviation and median (minimum-maximum) for numeric variables. Multiple logistic regression analysis will be used to estimate odds ratio for risk factors to development of AKI.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the ICU with a stay of 48 h or more

Exclusion Criteria:

* Patients with missing data, end-stage renal disease, existence of AKI at the time of ICU admission or history of renal transplantation will be excluded from the study. Patients that were readmitted to the ICU within 48 h will reunited with the first admission and be considered as one admission for the analysis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who developed acute kidney inhury during intensive care unit stay.
Sampling Method: Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-24 (Estimated); Study Completion 2023-11-24 (Estimated)

PRIMARY OUTCOMES:
To assess the incidence of acute kidney injury in ICU patients | Up to 28 day
  During their management lasting more than 48 hours in the ICU, some patients develop acute kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Uzman, Assoc. prof., Study Director — Health Science Unibersity, Haseki Training and Research Hospital
Locations (1):
- Health Science University, Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)